CLINICAL TRIAL: NCT00332371
Title: COMPACT (COMbining Plasma-filtration and Adsorption Clinical Trial): Efficacy and Safety of CPFA (Coupled Plasma Filtration Adsorption) for Septic Shock in the ICU
Brief Title: COMPACT - COMbining Plasma-filtration and Adsorption Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely interrupted for futility.
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Collaborators: Bellco Srl Mirandola, Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4817; ISRCTN24534559
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Shock, Septic
Keywords: Intensive Care; Shock, Septic; Adsorption; Sorption Detoxification
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Device: CPFA (Coupled Plasma Filtration Adsorption)
- 2 (No Intervention)

INTERVENTIONS:
Device: CPFA (Coupled Plasma Filtration Adsorption) — CPFA is a specific method for the treatment of sepsis.
  It consists of:
  1. a plasma-filter (polyethersulfone 0.45 m2 with a cutoff of approx 800 kDa)
  2. a hemofilter (polyethersulfone 1,4 m2)
  3. a cartridge (contains approximately 140 ml of hydrophobic styrenic resin)
  The kit is lodged in the Bellco "Lynda" machine (Bellco Mirandola, Italy). The treatment consists of the separation of plasma from the whole blood with adsorption of the inflammatory mediators and cytokines from the plasma, and a subsequent purification step by way of a hemofilter.
  Other Names: Coupled Plasma Filtration Adsorption
  Arms: 1

SUMMARY:
The study objective is to clarify whether the application of CPFA (coupled plasma-filtration adsorption) in addition to the current clinical practice is able to reduce mortality and prevent organ failures in septic shock patients in intensive care unit (ICU).

DETAILED DESCRIPTION:
Septic shock is a life-threatening clinical condition characterized by cardiovascular failure as a consequence of infection. Septic shock frequently causes multi-organ failure in the ICU. For this reason the extracorporeal therapies for the treatment of renal failure have become widespread in the ICU and, at the same time, new extracorporeal depurative techniques have been developed for the removal of inflammatory mediators. One of these techniques is CPFA (coupled plasma-filtration adsorption) that uses a sorbent once the separation between plasma and blood has been obtained with a plasma filter. The study objective is to clarify whether the application of CPFA in addition to the current clinical practice is able to reduce mortality and prevent organ failures in septic shock patients in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU in septic shock
* All patients that develop septic shock while in the ICU

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Cardiopulmonary resuscitation
* Cerebral coma
* Metastatic cancer
* Presence of relative or absolute contraindications to CPFA
* Estimated life expectancy less than 2 weeks
* Already included in the study
* Admission from an other ICU where the patient remained for more than 24 hours
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Hospital mortality (for patients discharged to other hospital, it will be intended as mortality at the discharge from the latest hospital in which the patients stayed) | At the discharge from the latest hospital

SECONDARY OUTCOMES:
Mortality within 90 days from randomization | 90 days from randomization
New organ failures (assessed through SOFA score) | Within ICU stay
Days not spent in the ICU during the first 30 days from randomization | 30 days from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Livigni, MD, Principal Investigator — Ospedale San Giovanni Bosco, Torino, ITALY
Locations (19):
- Italy (19):
  - Ospedale SS. Antonio e Biagio e C. Arrigo, Alessandria, AL
  - Ospedale Regionale della Valle d'Aosta, Servizio Anestesia e Rianimazione, Aosta, AO
  - Ospedali Riuniti, I Servizio Anestesia e Rianimazione, Bergamo, BG
  - Ospedale Policlinico San Pietro, Servizio Anestesia e Rianimazione, Ponte San Pietro, BG
  - Ospedale Policlinico San Marco, Terapia Intensiva, Zingonia, BG
  - Ospedale Spedali Civili, II Servizio di Anestesia e Rianimazione, Brescia, BS
  - Ospedale Vittorio Emanuele, II Servizio di Anestesia e Rianimazione, Catania, CT
  - Ospedale Morgagni-Pierantoni, U.O. Anestesia e Rianimazione, Forlì, FC
  - Ospedale Careggi - Villa Monna Tessa, TI Polifunzionale e Post-trapianto, Florence, FI
  - Ospedale S. Giovanni di Dio ASL 10, Servizio Anestesia e Rianimazione, Florence, FI
  - Ospedale Civile, Imperia, IM
  - Ospedale Civile, Servizio Anestesia e Rianimazione, Sanremo, IM
  - Ospedale A. Manzoni, U.O. Anestesia e Rianimazione 1, Lecco, LC
  - Ospedale Madonna delle Grazie, U.O. Anestesia e Rianimazione, Matera, MT
  - Ospedale di S. Chiara, VI U.O. di Anestesia, Rianimazione e Pronto Soccorso, Pisa, PI
  - European Hospital, Roma, RM
  - Ospedale San Camillo Forlanini, Roma, RM
  - Ospedale Civile Regione Piemonte ASL 9, Servizio Anestesia e Rianimazione, Ivrea, TO
  - Ospedale San Giovanni Bosco, Servizio Anestesia e Rianimazione B-DEA, Torino, TO

REFERENCES:
- [Derived] Livigni S, Bertolini G, Rossi C, Ferrari F, Giardino M, Pozzato M, Remuzzi G; GiViTI: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Italian Group for the Evaluation of Interventions in Intensive Care Medicine) is an independent collaboration network of Italian Intensive Care units. Efficacy of coupled plasma filtration adsorption (CPFA) in patients with septic shock: a multicenter randomised controlled clinical trial. BMJ Open. 2014 Jan 8;4(1):e003536. doi: 10.1136/bmjopen-2013-003536. PMID 24401721
- See also: GiViTI official web site — http://www.giviti.marionegri.it